CLINICAL TRIAL: NCT02813876
Title: Application of Surgical Enhanced Recovery Techniques in Acute Pancreatitis
Brief Title: Enhanced Recovery in Acute Pancreatitis
Acronym: ASERT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Bechien U. Wu, Center for Pancreatic Care, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 10920
Record Dates: First submitted 2016-06-23; First posted 2016-06-27 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced recovery (Experimental): Enhanced recovery protocol for nursing, diet and analgesic regimen
  Interventions: Other: Enhanced recovery protocol
- Standard care (No Intervention): Standard care arm

INTERVENTIONS:
Other: Enhanced recovery protocol
  Arms: Enhanced recovery

SUMMARY:
Prospective randomized-controlled trial evaluating impact of enhanced recovery protocol compared to standard care for recovery of patients with acute pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* Acute pancreatitis confirmed by clinical history, serologic testing and/or radiographic imaging

Exclusion Criteria:

* • Severe acute pancreatitis defined as the presence of any of the following:

  * Organ failure (oxygen saturation<90% on room air, mean arterial pressure<70 mmHG or any requirement for vasopressor or inotropic support, serum creatinine>2.0, Glasgow coma score<15)
  * Suspected or confirmed infected pancreatic necrosis: fever, leukocytosis in the setting of suspicious findings on cross-sectional imaging (gas within necrotic collection) or confirmed infection on fine needle aspirate

    * Chronic pancreatitis or any chronic pain syndrome requiring use of narcotic analgesic within 30 days prior to hospitalization
    * Abdominal surgery within 60 days prior to hospitalization
    * History of gastrointestinal motility disorder
    * Inflammatory bowel disease
    * Chronic comorbid illness including but not limited to >New York Heart Association Class II congestive heart failure, cirrhosis, oxygen-dependent chronic obstructive pulmonary disease or malignancy other than non-squamous skin cancer not in remission.
    * Documented allegy to any of the following medications: dilaudid, Tylenol
    * Patients transferred from an outside hospital for ongoing care
    * Non-English speaking patients for whom an appropriate language interpretor cannot be identified.
    * Pregnant women will be excluded from participation in this phase IIb trial given the limited projected sample size and rarity of this condition during pregnancy.
    * Minors (patients <18 years of age) will not be eligible for study inclusion. The interventions being compared in the study protocol are standard care for adult patients with acute pancreatitis. However, the safety and efficacy of these treatments in the pediatric population has not been established.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Time to tolerance of oral refeeding | Up to 7 days
  Resumption of intake of 50% of solid meal without symptoms of worsening post-prandial abdominal pain, nausea or vomiting

SECONDARY OUTCOMES:
Time to disease resolution | Up to 30 days
  Acute Pancreatitis Clinical Activity Index score<50
Satisfaction with inpatient hospital care | 30 days post-hospitalization
  Comparison of overall and pain management satisfaction score based on validated survey instrument

CONTACTS AND LOCATIONS:
Overall Officials: Bechien U Wu, MD, MPH, Principal Investigator — Kaiser Permanente Southern California, Los Angeles Medical Center
Locations (1):
- Kaiser Permanente Los Angeles Medical Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Dong E, Chang JI, Verma D, Butler RK, Villarin CK, Kwok KK, Chen W, Wu BU. Enhanced Recovery in Mild Acute Pancreatitis: A Randomized Controlled Trial. Pancreas. 2019 Feb;48(2):176-181. doi: 10.1097/MPA.0000000000001225. PMID 30629020